CLINICAL TRIAL: NCT05056233
Title: Systane Hydration in Subjects Undergoing Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DER646-P001
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye Disease; Cataract
MeSH Terms: conditions — Dry Eye Syndromes; Cataract

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systane Hydration (Experimental): Systane Hydration lubricant eye drops dosed 4 times a day for 6 weeks (2 weeks prior to surgery and 4 weeks post surgery), with investigator defined post-operative standard of care
  Interventions: Other: Systane Hydration lubricant eye drops
- No Treatment (No Intervention): Investigator defined post-operative standard of care

INTERVENTIONS:
Other: Systane Hydration lubricant eye drops — Sterile solution indicated for the temporary relief of burning and irritation due to dryness of the eye
  Other Names: Systane Hydration® Ophthalmic Solution
  Arms: Systane Hydration

SUMMARY:
The primary objective of this study is to demonstrate reduced corneal staining with use of Systane Hydration among subjects with dry eye disease (DED) undergoing routine cataract removal and monofocal intraocular lens (IOL) implantation.

DETAILED DESCRIPTION:
Subjects will attend 6 scheduled study visits for an individual duration of participation of 6 weeks. One eye (study eye) will be followed.

ELIGIBILITY:
Key Inclusion Criteria:

* Seeking routine (age-related) cataract extraction with monofocal intraocular lens implantation;
* Able to provide informed consent;
* Willing and able to attend all study visits and comply with treatment;
* Have dry eyes per dry eye questionnaire.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Subjects who use of ocular drugs, other than the test article (for treatment group only) and other standard of care postoperative medications, during the study;
* History of intraocular or corneal surgery in the study eye;
* Use of artificial tears, steroids, or other medications as specified in the protocol;
* Clinically significant corneal scarring;
* Corneal degeneration, retinal degeneration or other ocular pathology as specified in the protocol.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Corneal staining | Up to Day 30 post-operative
  The National Eye Institute (NEI) grading scale will be used to evaluate the five corneal regions: Superior, inferior, central, temporal and nasal. Each region will be graded on a 0-3 scale, where 0 = normal (no staining), 1 = mild/superficial stippling micropunctate staining, 2 = moderate/macropunctate staining with some coalescent areas, and 3 = severe/numerous coalescent macropunctate areas and/or patches. The regions will be summed for a resultant overall score of 0 to 15.

SECONDARY OUTCOMES:
DEQ-5 Score | Up to Day 30 post-operative
  The Dry Eye Questionnaire-5 (DEQ-5) is a patient-reported outcome measures questionnaire designed to assess symptoms of dry eye disease. Subjects will respond to 5 questions using a 0-4 Likert-type scale, for a resultant overall score of 0 (best) to 20 (worst).
Ocular Comfort Questionnaire Score: My eyes are comfortable | Up to Day 30 post-operative
  Subjects will provide a comfort score (strongly disagree, disagree, neither agree nor disagree, agree, strongly agree) to the following question: "My eyes are comfortable."
Ocular Comfort Questionnaire Score: At the end of the day, my eyes feel comfortable | Up to Day 30 post-operative
  Subjects will provide a comfort score (strongly disagree, disagree, neither agree nor disagree, agree, strongly agree) to the following question: "At the end of the day, my eyes feel comfortable."
Ocular Comfort Questionnaire Score: My eyes are comfortable all day long | Up to Day 30 post-operative
  Subjects will provide a comfort score (strongly disagree, disagree, neither agree nor disagree, agree, strongly agree) to the following question: "My eyes are comfortable all day long."

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Surgical, Study Director — Alcon Research, LLC
Locations (1):
- Principal Investigator, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No